CLINICAL TRIAL: NCT00536510
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Demonstrate the Lipid-Altering Efficacy and Safety and Tolerability of MK0524A in Patients With Primary Hypercholesterolemia or Mixed Hyperlipidemia
Brief Title: Effect of MK0524A on Cholesterol Levels (0524A-048)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0524A-048; 2007_621
Record Dates: First submitted 2007-09-26; First posted 2007-09-27 (Estimated); Results first posted 2009-05-13 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Hypercholesterolemia; Hyperlipidemia
Keywords: High Cholesterol; Excess lipids
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias | interventions — MK-0524; Niacin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): laropiprant/niacin (MK0524A)
  Interventions: Drug: laropiprant/niacin (MK0524A)
- 2 (Placebo Comparator): placebo
  Interventions: Drug: Comparator: placebo

INTERVENTIONS:
Drug: laropiprant/niacin (MK0524A) — Treatment Period 1: one 20mg/1g tablet laropiprant/niacin once daily for 4 weeks
  Treatment Period 2: two 20mg/1g tablets laropiprant/niacin once daily for 8 weeks.
  All patients will receive placebo for a 4 week run-in period before randomization
  Other Names: MK0524A
  Arms: 1
Drug: Comparator: placebo — Treatment Period 1: one 20mg/1g tablet placebo to laropiprant/niacin once daily for 4 weeks
  Treatment Period 2: two 20mg/1g tablets of placebo to laropiprant/niacin once daily for 8 weeks.
  All patients will receive placebo for a 4 week run-in period before randomization.
  Arms: 2

SUMMARY:
The primary objective of the study is to assess the effects of MK0524A in reducing cholesterol levels in an Asian population.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female between 18 and 70 years of age
* Females of reproductive potential must agree to take acceptable contraceptive precautions for the duration of the study

Exclusion Criteria:

* Patient has a history of not being able to take niacin or niacin-containing products
* Patient consumes more than 2 alcoholic beverages per day
* Patient has poorly controlled Type 1 or Type 2 diabetes mellitus
* Patient engages in vigorous exercise or an aggressive diet regimen

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 646 (Actual)
Dates: Start 2007-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Kush D, Kim HS, Hu DY, Liu J, Sirah W, Sapre A, McCrary Sisk C, Paolini JF, Maccubbin D. Lipid-modifying efficacy of extended release niacin/laropiprant in Asian patients with primary hypercholesterolemia or mixed hyperlipidemia. J Clin Lipidol. 2009 May-Jun;3(3):179-86. doi: 10.1016/j.jacl.2009.04.048. Epub 2009 May 3. PMID 21291812

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase III
  First Patient In: 10-May-2007
  Last Patient Last Visit: 11-Mar-2008
  42 Outpatient centers in China (21), Hong Kong (2), India (11), and Korea (8)
Pre-assignment Details: Asia-regional lipid study with patients 18-70 yrs, including diabetic patients +/- statin, without ischemic vascular disease and LDL-C<130 mg/dL (3.37 mmol/L), patients on a statin with ≥2 risk factors with LDL-C ≥130 and ≤160 mg/dL (3.37 and 4.14 mmol/L), and patients +/- statin with ≤1 risk factor with ≥130 and ≤190 mg/dL (3.37 and 4.92 mmol/L).
Groups:
- MK0524A 2 g: All patients received placebo for a 4 week run-in period before randomization.
  Drug: laropiprant/niacin (MK0524A)
  Treatment Period 1: one 20 mg /1 g tablet of laropiprant/niacin once daily for 4 weeks.
  Treatment Period 2: two 20 mg /1 g tablets of laropiprant/niacin once daily for 8 weeks.
- Placebo: All patients received placebo for a 4 week run-in period before randomization.
  Drug: Comparator: placebo
  Treatment Period 1: one 20 mg /1 g tablet placebo to laropiprant/niacin once daily for 4 weeks
  Treatment Period 2: two 20 mg /1 g tablets of placebo to laropiprant/niacin once daily for 8 weeks.
Period: Overall Study
Arm/Group | MK0524A 2 g | Placebo
Started | 322 | 324
Completed | 240 | 295
Not Completed | 82 | 29
Not completed — Adverse Event | 27 | 4
Not completed — Lost to Follow-up | 11 | 8
Not completed — Protocol Violation | 4 | 5
Not completed — Withdrawal by Subject | 16 | 9
Not completed — Flushing with Product | 20 | 0
Not completed — Laboratory Adverse Event | 2 | 1
Not completed — Patient Discontinued for Other Reasons | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK0524A 2 g | Placebo | Total
Number analyzed (Participants) | 322 | 324 | 646
Age, Customized [Number; unit: participants]
  <65 years | 276 | 279 | 555
  >=65 years | 46 | 45 | 91
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 191 | 185 | 376
  Male | 131 | 139 | 270
Concomitant Statin Use [Number; unit: Participants]
  Yes | 150 | 146 | 296
  No | 172 | 178 | 350
Country [Number; unit: Participants]
  China (includes Hong Kong) | 159 | 158 | 317
  India | 82 | 79 | 161
  Korea | 81 | 87 | 168
Glycemic Status [Number; unit: Participants] — Fasting Plasma Glucose (FPG)
  *Glycemic Status (Source: American Diabetes Association Guidelines)
  * Normal - FPG level of less than 100 mg/dL
  * Impaired Glucose - FPG level between 100 & 125 mg/dL
  * Diabetic - FPG level of 126 mg/dL or higher
  Participants
    Normal* | 166 | 156 | 322
    Impaired Glucose* | 8 | 4 | 12
    Diabetic* | 148 | 164 | 312
High Density Lipoprotein Cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 48.1 (10.8) | 48.5 (11.8) | 48.3 (11.3)
Low Density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] | 124 (34.4) | 121.8 (34.0) | 122.9 (34.2)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) After 12 Weeks
Description: Low Density Lipoprotein Cholesterol (LDL-C) after 12 weeks is calculated as the difference between week 12 measure and baseline measure divided by baseline measure *100
Time Frame: 12 weeks
Population: Full Analysis Set: consisted of all randomized patients who (i) took at least one dose of the treatment period study medication and (ii) had a baseline measurement and at least one measurement during Weeks 5 to 12. The last available lipid values during Weeks 5 to 12 were used for patients who had no lipid data collected at Week 12.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | MK0524A 2 g | Placebo
Number analyzed (Participants) | 259 | 298
Percent Change | -10.3 [-13.2 to -7.4] | 4.4 [1.7 to 7.2]
Statistical Analysis 1: Comparison: MK0524A 2 g vs Placebo; The primary hypothesis of superiority of MK0524A 2 g to placebo in lowering Low Density Lipoprotein Cholesterol (LDL-C) was assessed using the comparison between these 2 groups from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — The significance test was 2-tailed with α=0.05; The efficacy analysis was performed using an ANOVA model with factors for treatment, country, gender, and stratum defined by concomitant statin use; Mean Difference (Final Values) = -14.7, 95% CI [-18.6 to -10.9], Standard Error of Mean 1.96

2. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C) After 12 Weeks
Description: Percent change from baseline in High Density Lipoprotein Cholesterol (HDL-C) after 12 weeks is calculated as the difference between week 12 measure and baseline measure divided by baseline measure *100
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | MK0524A 2 g | Placebo
Number analyzed (Participants) | 259 | 300
Percent Change | 18.6 [16.1 to 21.1] | 2.6 [0.3 to 5.0]
Statistical Analysis 1: Comparison: MK0524A 2 g vs Placebo; The secondary hypothesis of superiority of MK0524A 2 g to placebo in lowering High Density Lipoprotein Cholesterol (HDL-C) was assessed using the comparison between these 2 groups from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — The significance test was 2-tailed with α=0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 15.9, 95% CI [12.6 to 19.2], Standard Error of Mean 1.68

ADVERSE EVENTS:
Description: The number of participants at risk for laboratory adverse events represents participants for whom laboratory test results were recorded postbaseline.
Arm/Group | MK0524A 2 g | Placebo
Serious Adverse Events (participants affected / at risk) | 3/321 | 2/323
Other Adverse Events (participants affected / at risk) | 123/321 | 54/323
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK0524A 2 g (N=321) | Placebo (N=323)
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis Haemorrhagic (Gastrointestinal disorders) | 1 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint Injury (Injury, poisoning and procedural complications) | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | MK0524A 2 g (N=321) | Placebo (N=323)
Nausea (Gastrointestinal disorders) | 10 | 5
Upper Respiratory Tract Infection (Infections and infestations) | 7 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 26 | 3
Rash (Skin and subcutaneous tissue disorders) | 13 | 2
Flushing (Vascular disorders) | 37 | 8
Alanine Aminotransferase Increased (Endocrine disorders) | 9/298 | 9/310
Creatine Phosphokinase Increased (Endocrine disorders) | 12/299 | 9/310
Fasting Blood Glucose Increased (General disorders) | 9/281 | 7/302
Protein Urine Present (Renal and urinary disorders) | 1/33 | 1/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.